CLINICAL TRIAL: NCT04152642
Title: A Pilot Clinical Study to Assess Dry Mouth Relief After Using an Experimental Mouth Rinse Compared to a Negative Control
Brief Title: A Pilot Study to Assess Dry Mouth Relief After Using an Experimental Mouth Rinse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Procter and Gamble (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CSD2019138
Record Dates: First submitted 2019-11-01; First posted 2019-11-05 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Dry Mouth
MeSH Terms: conditions — Xerostomia

STUDY DESIGN:
Intervention Model Description: 3-treatment crossover, with 4 days of use
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Marketed Mouth Rinse (Active Comparator): dry mouth rinse to be taken up to 5x a day, at least twice a day, 15 ml for 30 seconds. Subjects will be restricted from using mouth rinse, acclimation products, eating or drinking for 4-hours after first use (on-site) on Day 1 and Day 4.
  Interventions: Device: Marketed Dry Mouth Rinse
- Experimental Mouth Rinse (Experimental): dry mouth rinse to be taken up to 5x a day, at least twice a day, 15 ml for 30 seconds. Subjects will be restricted from using mouth rinse, acclimation products, eating or drinking for 4-hours after first use (on-site) on Day 1 and Day 4.
  Interventions: Device: Experimental Dry Mouth Rinse
- Water/Negative Control (Sham Comparator): subjects will swallow 15 ml of water (on-site). Subjects will be restricted from using mouth rinse, acclimation products, eating or drinking for 4-hours after water intake (on-site) on Day 1 and Day 4.
  Interventions: Other: Water control

INTERVENTIONS:
Device: Marketed Dry Mouth Rinse — relieves dry mouth symptoms by physically coating oral mucosal surfaces.
  Arms: Marketed Mouth Rinse
Other: Water control — negative control
  Arms: Water/Negative Control
Device: Experimental Dry Mouth Rinse — relieves dry mouth symptoms by physically coating oral mucosal surfaces.
  Arms: Experimental Mouth Rinse

SUMMARY:
The objective of this pilot study is to determine if an experimental mouth rinse and a marketed dry mouth rinse are more effective in relieving dry mouth compared to water.

DETAILED DESCRIPTION:
This is a controlled, randomized, 3-treatment, 3-period crossover study in subjects with self-reported dry mouth symptoms as determined by subject responses (as determined by the response to "relieving the discomfort of dry mouth" question from the modified Product Performance and Attributes Questionnaire I/ Moisturization and Dryness (PPAQ I/ MD)) compared to water. Subjects enrollment is based on the responses to the Dry Mouth Inventory (DMI). A sufficient number of volunteers will be screened to ensure enrollment of up to 30 subjects at Acclimation. Subjects who meet the eligibility criteria will continue into the treatment phase of the study. Safety will be assessed by Oral examinations at Baseline/Day1 and Day 4. Subjects will complete questionnaires at Baseline (before product use Day 1 only), after immediate use, 30 minutes, 1 hour, 2 hours, and 4 hours after supervised product use on Day 1 and Day 4 of each period. The PPAQ II questionnaire will be completed in the morning of Day 4 of each period. Subjects will be randomly assigned to treatment sequences at the Baseline visit of Period 1. The treatment and washout periods will be repeated until all three treatment periods have been completed.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent prior to participation and be given a signed copy of the informed consent form;
* Be at least 18 years of age;
* Be in good general health as determined by the Investigator/designee;
* Agree not to participate in any other oral care studies for the duration of this study;
* Agree to delay elective dentistry, including dental prophylaxis, until study completion, and to report any non-study dentistry received during the course of the study;
* Agree to refrain from the use of any non-study oral hygiene products for the study duration including mouth rinse and toothpaste (flossing is permitted if part of their normal routine);
* Self-report a dry mouth feeling according to the modified DMI questions. (Subject must answer at least 2 out of 4 questions with 'agree a little,' 'agree' or 'strongly agree');
* Agree to refrain from smoking, drinking, using tobacco products, using breath mints, medicated lozenges, or chewing gum during the 4-hour test period;
* Agree to return for all scheduled visits and to follow all study procedures.

Exclusion Criteria:

* Any condition or disease, as determined by the Investigator/Designee, that could be expected to interfere with examination procedures, with compliance, or with the subject's safe completion of the study;
* Severe periodontal disease, as characterized by purulent exudate, generalized mobility, and/or severe recession;
* Active treatment for periodontitis;
* Having a history of allergies or hypersensitivity to mouth rinse or ingredients in commercial dental products or cosmetics;
* Self-reported pregnancy or the intent to become pregnant during the study, or breast feeding;
* Full or partial dentures or any orthodontic appliances such as braces or aligners, or tongue or mouth piercing;
* Having diabetes;
* Inability to undergo any study procedure;
* Having untreated oral mucosal disease which in the opinion of the investigator could interfere with the study (e.g., current oral ulceration);
* Use of prescription systemic parasympathetic medications (e.g., Pilocarpine), for the treatment of the feeling of dry mouth;
* Currently under the care of a dental/medical professional specifically for the treatment of dry mouth (at the discretion of the Investigator/Designee);
* Self-reported mouth breathers (i.e., mouth breathing secondary to nasal obstruction);
* Evidence of gross intra-oral neglect or need for extensive dental therapy; or
* Currently undergoing radiotherapy and/or chemotherapy treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-11-04 (Actual); Primary Completion 2019-12-05 (Actual); Study Completion 2019-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Malgorzata Klukowska, DDS, Principal Investigator — Procter and Gamble
Locations (1):
- Procter & Gamble, Mason, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects that qualified were randomized to one of six treatment sequences: ABC, ACB, BCA, BAC, CAB, or CBA. Subjects had at least a 3 day washout before Period 1 and in-between each period.
Groups:
- Overall Study: Single-center, randomized 3-treatment, 3-periods cross-over study.
Period: Overall Study
Arm/Group | Overall Study
Started | 22
C (Water/Negative) Control (This was a 3-treatment, 3-period, cross-over design. Each subject was assigned to receive each treatment. Each period lasted 4 days.) | 20
A (Marketed Rinse) (This was a 3-treatment, 3-period, cross-over design. Each subject was assigned to receive each treatment. Each period lasted 4 days.) | 19
B (Experimental Rinse) (This was a 3-treatment, 3-period, cross-over design. Each subject was assigned to receive each treatment. Each period lasted 4 days.) | 19
Completed (15 subjects received all 3 treatment products) | 15
Not Completed | 7

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: single-center, randomized 3-treatment, 3-period crossover study
Arm/Group | Overall Study
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (11.96)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Dry Mouth Inventory [Count of Participants; unit: Participants] — subjects had to answer 2 of the 4 dry mouth inventory questions positively. How much do you agree or disagree that you experience the following? (strongly disagree, disagree, disagree a little, agree a little, agree, strongly agree)
  1. No moisture in the mouth
  2. Lips sticking to teeth
  3. Tongue sticking to roof of mouth
  4. Throat feels dry
  Participants
    No moisture in the mouth: Agree a Little, Agree, or Strongly Agree | 19
    No moisture in the mouth: Disagree a Little, Disagree, or Strongly Disagree | 3
    Lips sticking to teeth: Agree a Little, Agree, or Strongly Agree | 18
    Lips sticking to teeth: Disagree a Little, Disagree, or Strongly Disagree | 4
    Tongue sticking to roof of mouth: Agree a Little, Agree, or Strongly Agree | 13
    Tongue sticking to roof of mouth: Disagree a Little, Disagree, or Strongly Disagree | 9
    Throat feels dry: Agree a Little, Agree, or Strongly Agree | 22
    Throat feels dry: Disagree a Little, Disagree, or Strongly Disagree | 0

OUTCOME MEASURES:

1. Primary Outcome: Product Performance and Attributes (PPAQ I) Question #1: 2-hr at Day 4
Description: Product Performance and Attributes (PPAQ I) Question #1:
  Since you have been used the product, please rate each of the following at this timepoint: (Select one response for each attribute)- excellent=5, very good=4, good=3, fair=2, poor=1:
  1) Relieves the discomfort of your dry mouth
Time Frame: 2-hour, Day 4
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Water/Negative Control | Marketed Mouth Rinse | Experimental Mouth Rinse
Number analyzed (Participants) | 20 | 19 | 19
units on a scale | 1.79 (0.197) | 2.97 (0.204) | 3.33 (0.203)

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the entire duration of the study for each intervention, an average of 1 month.
Arm/Group | Water/Negative Control | Marketed Mouth Rinse | Experimental Mouth Rinse
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/19 | 0/19
Other Adverse Events (participants affected / at risk) | 5/20 | 3/19 | 2/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Water/Negative Control (N=20) | Marketed Mouth Rinse (N=19) | Experimental Mouth Rinse (N=19)
Stomatitis (Gastrointestinal disorders) | 3 | 1 | 1
mouth injury (Injury, poisoning and procedural complications) | 1 | 1 | 0
oral herpes (Infections and infestations) | 1 | 0 | 0
cheilitis (Gastrointestinal disorders) | 0 | 0 | 1
Gingival Pain (Gastrointestinal disorders) | 0 | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/42/NCT04152642/Prot_SAP_001.pdf